CLINICAL TRIAL: NCT05242861
Title: A Retrospective Study of Brachytherapy in Gynecological Cancers
Brief Title: Retrospective Study of Brachytherapy
Acronym: RetroBT
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BTOG 2201
Record Dates: First submitted 2022-02-06; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Brachytherapy; Uterine Cervical Neoplasms; Uterine Neoplasms; Vulvar Cancer; Vaginal Cancer; Ovarian Neoplasms; Gynecologic Neoplasm
Keywords: Brachytherapy; Cervical Cancer; Endometrial Cancer; Vaginal Cancer; Vulvar Cancer; Image Guided; 3D Print
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Ovarian Neoplasms; Genital Neoplasms, Female; Endometrial Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cervix radical BT
  Interventions: Radiation: Brachytherapy
- Cervix adjuvant BT
  Interventions: Radiation: Brachytherapy
- Cervix palliative BT
  Interventions: Radiation: Brachytherapy
- Uterus BT
  Interventions: Radiation: Brachytherapy
- Other GO cancer BT
  Interventions: Radiation: Brachytherapy

INTERVENTIONS:
Radiation: Brachytherapy — Applicator, dose, schedule, technology, image, 3D print, efficacy, toxicity of brachytherapy

SUMMARY:
Brachytherapy for gynecological cancers will be studied retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 80 female
* Underwent brachytherapy
* With gynecological cancer

Exclusion Criteria:

* Refusal to enter this trial

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 to 80 years old female who diagnosed as gynecological cancer and underwent brachytherapy will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 5-year
  the percentage of participants in the group who survives

SECONDARY OUTCOMES:
Progression-free survival rate | 5-year
  the percentage of participants in the group whose disease is likely to remain stable
Side effects | 5-year
  side effects associated with treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Sturdza A, Potter R, Fokdal LU, Haie-Meder C, Tan LT, Mazeron R, Petric P, Segedin B, Jurgenliemk-Schulz IM, Nomden C, Gillham C, McArdle O, Van Limbergen E, Janssen H, Hoskin P, Lowe G, Tharavichitkul E, Villafranca E, Mahantshetty U, Georg P, Kirchheiner K, Kirisits C, Tanderup K, Lindegaard JC. Image guided brachytherapy in locally advanced cervical cancer: Improved pelvic control and survival in RetroEMBRACE, a multicenter cohort study. Radiother Oncol. 2016 Sep;120(3):428-433. doi: 10.1016/j.radonc.2016.03.011. Epub 2016 Apr 29. PMID 27134181
- [Background] Lindegaard JC, Madsen ML, Traberg A, Meisner B, Nielsen SK, Tanderup K, Spejlborg H, Fokdal LU, Norrevang O. Individualised 3D printed vaginal template for MRI guided brachytherapy in locally advanced cervical cancer. Radiother Oncol. 2016 Jan;118(1):173-5. doi: 10.1016/j.radonc.2015.12.012. Epub 2015 Dec 29. PMID 26743833
- [Background] Sekii S, Tsujino K, Kosaka K, Yamaguchi S, Kubota H, Matsumoto Y, Ota Y, Sasaki R, Soejima T. Inversely designed, 3D-printed personalized template-guided interstitial brachytherapy for vaginal tumors. J Contemp Brachytherapy. 2018 Oct;10(5):470-477. doi: 10.5114/jcb.2018.78832. Epub 2018 Oct 9. PMID 30479625
- [Background] Harris BD, Nilsson S, Poole CM. A feasibility study for using ABS plastic and a low-cost 3D printer for patient-specific brachytherapy mould design. Australas Phys Eng Sci Med. 2015 Sep;38(3):399-412. doi: 10.1007/s13246-015-0356-3. Epub 2015 Jun 25. PMID 26108891
- [Result] Han K, Milosevic M, Fyles A, Pintilie M, Viswanathan AN. Trends in the utilization of brachytherapy in cervical cancer in the United States. Int J Radiat Oncol Biol Phys. 2013 Sep 1;87(1):111-9. doi: 10.1016/j.ijrobp.2013.05.033. Epub 2013 Jul 9. PMID 23849695